CLINICAL TRIAL: NCT04189302
Title: Comparative Evaluation of Two Surgical Blade Designs to Harvest Palatal Connective Tissue Graft by Single Incision Technique: A Randomized Controlled Clinical Trial
Brief Title: Comparative Evaluation of Two Surgical Blades
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Krishnadevaraya College of Dental Sciences & Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 02_D012_101317
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Wound Healing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- palatal connective tissue graft harvest with KPM blade (Experimental): palatal connective tissue graft is harvested using single incision technique using KPM blade
  Interventions: Procedure: connective tissue graft harvest using KPM blade
- palatal connective tissue graft harvest with 15C blade (Active Comparator): palatal connective tissue graft is harvested using single incision technique using 15 C blade
  Interventions: Procedure: connective tissue graft harvest using 15 C blade

INTERVENTIONS:
Procedure: connective tissue graft harvest using KPM blade — after local anesthesia is injected, the surgical procedure is initiated with 15 C blade and the connective tissue graft is detached from epithelium and underlying periosteum. then the connective tissue is harvested with the help of 2 vertical and 1 horizontal incisions using KPM blade.
  Arms: palatal connective tissue graft harvest with KPM blade
Procedure: connective tissue graft harvest using 15 C blade — after local anesthesia is injected, the surgical procedure is initiated with 15 C blade and the connective tissue graft is detached from epithelium and underlying periosteum. then the connective tissue is harvested with the help of 2 vertical and 1 horizontal incisions using 15C blade.
  Arms: palatal connective tissue graft harvest with 15C blade

SUMMARY:
this study compares the ease of execution, wound healing and patient morbidity of 2 surgical blade designs.

DETAILED DESCRIPTION:
Over the past few years, connective tissue graft (CTG) is considered as a gold standard and reliable treatment modality in periodontal aesthetic surgeries.Various CTG harvesting techniques have been described which differ in the number of the incisions, flap design, and the technique for gaining access to the graft. Among the numerous techniques for CTG harvest, single incision technique (SIT) proposed by Hurzeler is described as more conservative and least traumatic for the patient. However, there are few limitations of SIT.

To overcome these difficulties, Kumar proposed a special instrument, Barraquer cataract knife and AVS blade to harvest CTG using modified SIT. The Barraquer cataract knife is an ophthalmic blade which is extremely thin and useful in giving mesial and distal incisions of CTG within the limited space under partial thickness flap without tearing it. AVS blade has a terminal shank angled at 100 degrees, with the smooth outer surface and the cutting edge at terminal end perpendicular to the long axis of the instrument which enables placement of medial incision easily without damaging the overlying flap. However, their proposed instrument too had limitations like need for two instruments to, and the straight angulation of the shank makes the adaptation difficult to the palatal vault.

A new instrument KPM blade has been envisaged eliminating these limitations. It has a long thin handle with two contra-angulations of 45degrees and 90degrees on the shank and a terminal shank of ten mm length.This makes the shank easily adapt to any form of the palatal vault, offsets the interference of palatal surfaces of molars and provides a depth control of ten mm in apico-coronal direction without causing any vascular troubles. From the terminal shank blade has a perpendicular projection of two mm which is curved and bevelled which enables it to be used in multidirection with better visibility and good clinical control on incision.

However, till date, this novel KPM blade has not been explored in harvesting CTG using SIT. Thus, the purpose of the present study is to compare KPM blade v/s standard 15c blade to harvest CTG in SIT in terms of ease of harvesting (time), early healing in palatal donor area and patient morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study.
2. Patients between age group of 25 to 55 years.
3. Systemically healthy subjects.
4. Patients with esthetic concerns.
5. Patients with palatal mucosa thickness greater than 2.5mm.
6. Full mouth plaque score (FMPS) < 20%, Full mouth bleeding score (FMBS) < 20%.

Exclusion Criteria:

1. Patients with any systemic diseases.
2. Patients with history of coagulation disorders.
3. Patients with immunological disorders.
4. Pregnant and lactating females.
5. History of tobacco usage in any form.
6. Patients taking medication that interfere with healing.
7. Patients with palatal mucosa thickness lesser than 2.5mm.
8. Patients who have undergone periodontal surgery within 6 months from the time they enrolled in the study.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-01 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
ease of execution | 1 month
  it is measured as a time parameter, where the surgical time taken is measured with stop watch
patient morbidity and postoperative course | 1 month
  a questionnaire will be given to the patients in which their responses for Visual Analog Score that ranges from 1-10 values and highest values indicate the worst outcome, variation in feeding habits, analgesics dosage is recorded. And during baseline and subsequent followups epithelization and bleeding are noted

SECONDARY OUTCOMES:
wound healing | 1 month
  wound healing at palatal donor site is evaluated using modified wound healing index

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Karthikeyan B.V, MDS, Principal Investigator — Krishnadevaraya college of dental sciences , Bangalore ,KARNATAKA , INDIA

IPD SHARING:
Plan to Share IPD: No